CLINICAL TRIAL: NCT00230022
Title: Pilot Clinical Trial of Computer-based Motivational Intervention
Brief Title: Pilot Clinical Trial of Computer-based Motivational Intervention - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-14621-1; R21DA014621 (NIH)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief computer-delivered intervention (Experimental): A 20-minute interaction with software designed to partially replicate the experience of a brief motivational intervention with a therapist or health care professional. Included decisional balance, normed feedback, and optional goal-setting.
  Interventions: Behavioral: Brief computer-delivered intervention
- Assessment only (No Intervention): Participants in this arm only completed assessment section, same as intervention group, but then was done.

INTERVENTIONS:
Behavioral: Brief computer-delivered intervention — 20-minute interaction with voice-enabled software that could provide reflections, images, text, etc.
  Arms: Brief computer-delivered intervention

SUMMARY:
Pilot trial of computer-based motivational intervention. Hypothesis: The brief computer-delivered intervention would result in higher motivation to change at follow-up.

DETAILED DESCRIPTION:
Participants were randomized into brief intervention vs. assessment-only conditions, with follow-up to measure overall motivation to change.

ELIGIBILITY:
Woman in immediate post-partum period

Inclusion Criteria:

Self-report of drug use prior to pregnancy

Exclusion Criteria:

Frank psychosis or other cognitive impairment; inability to communicate in English; fatigue; recent receipt of narcotic pain medication; grieving over medically compromised infant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, Ph.D., Principal Investigator — ACT
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Result] Ondersma SJ, Chase SK, Svikis DS, Schuster CR. Computer-based brief motivational intervention for perinatal drug use. J Subst Abuse Treat. 2005 Jun;28(4):305-12. doi: 10.1016/j.jsat.2005.02.004. PMID 15925264

RESULTS

PARTICIPANT FLOW:
Groups:
- Brief Computer-delivered Motivational Intervention: Brief computer-delivered intervention in three components: decisional balance, feedback, and optional goal setting.
- Assessment Only: Only assessment, same as completed by intervention group. No further interaction with computer.
Period: Overall Study
Arm/Group | Brief Computer-delivered Motivational Intervention | Assessment Only
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Computer-delivered Motivational Intervention | Assessment Only | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Baseline motivation [Mean (Standard Deviation); unit: units on a scale] — Visual analog scale questions were used to assess baseline motivation, self-efficacy, problem recognition, and change likelihood. The average of the items were calculated for baseline measurement resulting in a score ranging from 1 to 100. Higher scores represent increase motivation for change, self-efficacy, problem recognition and increased likelihood of making a change.
  units on a scale | 82.5 (18.9) | 79.5 (21.2) | 81.0 (20.3)

OUTCOME MEASURES:

1. Primary Outcome: Motivation to Change Substance Use
Description: An eight-item measure tapping motivation to change, self-efficacy, and change intention was assessed using visual analog scales. The average of the eight items was calculated resulting in a score ranging from 1 to 100. The measure was asked at baseline (reported in baseline data) and the one month follow-up. Scores here represent average level of motivation for change at the time of follow-up. Higher scores represent higher levels of motivation to change, self-efficacy and intention to change.
Time Frame: One month
Population: A total of 30 participants were included in this pilot trial, based primarily on convenience and timeframe. The primary goal was effect-size estimation, so power was not a primary concern. Last Observation Carried Forward(LOCF) was utilized for 8 participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Brief Computer-delivered Motivational Intervention: A brief assessment, plus a brief (20-minute) motivational intervention delivered solely by computer. The software was synchronously interactive and followed a traditional motivational interviewing approach.
- Assessment Only: Only assessment measures with no subsequent intervention.
Arm/Group | Brief Computer-delivered Motivational Intervention | Assessment Only
Number analyzed (Participants) | 15 | 15
units on a scale | 88.8 (10) | 77.4 (20)

ADVERSE EVENTS:
Arm/Group | Brief Computer-delivered Motivational Intervention | Assessment Only
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Small sample size in the pilot clinical trial. Because of this lack of power, a statistically significant difference between groups was not demonstrated, and the 95% Confidence Interval (CI) for the effect size estimate included zero.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No